CLINICAL TRIAL: NCT03379363
Title: Retrospective Chart Review Study of Pediatric Patients Treated With Korlym for Cushing Syndrome
Status: Terminated | Type: Observational
Why Stopped: Insufficient number of patients
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: C1073-900
Record Dates: First submitted 2017-10-24; First posted 2017-12-20 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Hypercortisolism; Cushing Syndrome
Keywords: cushing syndrome, hypercortisolism
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Cushing Syndrome Patients: Pediatrics patients with endogenous Cushing syndrome who received at least one dose of Korlym

SUMMARY:
This retrospective, multi-center, chart review study will collect patient data from medical charts of pediatric patients who have been treated with Korlym for Cushing's syndrome.

DETAILED DESCRIPTION:
This retrospective chart review study seeks to collect data from pediatric patients treated with Korlym (mifepristone) to help provide clinicians with some insight on the potential role of mifepristone in the treatment of pediatric patients with Cushing syndrome.

Only sites that have been identified to have patients appropriate for this protocol will be invited to participate and contribute data on their patients

Data to be collected from a retrospective chart review will include:

* Patient demographics
* Medical history
* Pre and post treatment clinical assessments and laboratory results
* Radiologic findings (if available)
* Adverse events

Data will be collected for all follow-up visits, up until the most recent encounter prior to IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics (age≤21 years) at time Korlym initiation
* Considered to have a diagnosis of endogenous Cushing's syndrome by the healthcare provider
* Received at least one dose of Korlym
* Availability of pre-treatment (baseline) and follow-up data

Exclusion Criteria:

* None

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients who have been treated with Korlym for Cushing's syndrome
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Drug utilization patterns as assessed by chart review | Length of Korlym therapy, up to 5 years
  The retrospective review would analyze the drug utilization patterns of pediatric patients treated with Korlym

SECONDARY OUTCOMES:
Weight as assessed by chart review | Length of Korlym therapy, up to 5 years
  The retrospective review would analyze changes in Weight (in kg) in pediatric patients treated with Korlym
Blood Pressure as assessed by chart review | Length of Korlym therapy, up to 5 years
  The retrospective review would analyze changes in Blood Pressure (in mmHg) in pediatric patients treated with Korlym

CONTACTS AND LOCATIONS:
Locations (1):
- Corcept Therapeutics, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: No